CLINICAL TRIAL: NCT04766879
Title: A Cluster Randomized Trial of the Efficacy of a Spatial Repellent (the Envelope) on Plasmodium Falciparum Malaria Incidence as Measured by Time to First Infection in Western Kenya
Brief Title: Spatial Repellents for the Prevention of Malaria in Kenya
Acronym: AEGIS Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: S.C. Johnson & Son, Inc. (Industry); Kenya Medical Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); fhiClinical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-08-5506
Record Dates: First submitted 2021-02-08; First posted 2021-02-23 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Malaria
Keywords: Malaria; Spatial Repellent; Transfluthrin; Vector-borne diseases; Mosquito vectors; Incidence
MeSH Terms: conditions — Malaria; Vector Borne Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spatial Repellent (Experimental): Transfluthrin
  Interventions: Device: Transfluthrin
- Placebo (Placebo Comparator): Inert ingredients
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Transfluthrin — Passive emanator with formulated transfluthrin
  Arms: Spatial Repellent
Device: Placebo — Passive emanator with formulated inert ingredients
  Arms: Placebo

SUMMARY:
Spatial repellents are chemical-based devices that when placed in a room, make that room non-conducive for mosquitoes. These tools can be used to help in the fight against vector borne diseases such as malaria and dengue. However, their efficacy in reducing mosquito biting and therefore malaria transmission has never been evaluated in Africa. This study will evaluate the efficacy of a spatial repellent in reducing mosquito biting on human beings and measure the impact any reduced biting will have on malaria transmission. The investigators will recruit and follow-up 5,984 children between 6 months and <10 years of age in Busia County to determine how many times they will be infected with malaria in villages where the investigators will have distributed spatial repellents and compare the rate of infection to villages where the investigators will not have distributed the repellent devices. Additionally, the investigators will measure whether the distribution of spatial repellents in one village will drive mosquitoes to their neighboring houses thereby increasing malaria transmission in those areas. The children participating in the study will be divided into 3 groups (cohorts). The first group will be followed up during the first 4 months before any intervention is distributed and the purpose here will be to determine that the villages are comparable. After this, the investigators will recruit the next group of participants and follow them up for 1 year and repeat this again for another year. During the follow-up, the children will be asked to come to the health facility where they will be tested for malaria using RDT or blood slide for microscopy. Every two weeks, a member of the study team will come to the participant's house and ask them if they had any history of fever. If the participants had fever, they will be tested for malaria. All children who turn out to be positive for malaria by RDT will be treated free of charge. At the same time, the investigators shall also perform mosquito collections to determine the impact of spatial repellents on the density of Anopheles mosquitoes.

DETAILED DESCRIPTION:
Spatial repellents (SRs) have been widely used for the prevention of mosquito bites but their protective efficacy (PE) in reducing mosquito-borne diseases has never been evaluated in Africa. To address this knowledge gap, western Kenya was selected as a site to estimate the impact of a transfluthrin-based spatial repellent on malaria-related outcomes in Busia County, where baseline malaria transmission ranges from 2.5 to 4.1 new infections per person per year.

A total of 5,984 children between 6 months and <10 years of age will be enrolled in three separate cohorts (baseline, cohort 1 and cohort 2). A total of 2,040 children from among 60 clusters will be enrolled for a four-month baseline prior to placement of the SR intervention. After baseline, a total of 1,972 participants from among 58 clusters, will be enrolled into cohort 1 and followed for one year. Cohort 2, consisting of a total of 1,972 children, will be enrolled from among 58 clusters to provide a total of two years of follow up. Children who have been selected for inclusion in the baseline cohort will be eligible for selection to cohort 1 or 2 but not both.

Cohort 1 and Cohort 2 during intervention will be split into two groups, one to estimate the direct effect of the SR (total of 1,624 children, 812 per follow up year) and a second to estimate the degree of diversion (or mass effect) of mosquitoes and malaria transmission from persons protected by the SR to persons who are unprotected (total of 2,320 children, 1,160 per follow up year). All cohorts will be followed once every two weeks with finger prick blood samples taken once every 4 weeks to test for malaria or whenever a participant reports a recent (within 48 hours) history of fever.

The incidence of malaria in the baseline cohort will be used to validate underlying assumptions prior to intervention. The incidence of malaria in each cohort followed with intervention will be estimated and compared to determine the benefit of using an SR in an area with high, year-round transmission of malaria. Monthly collections of mosquitoes using CDC light traps will be conducted to determine if there are entomological correlates of SR efficacy that may be useful for the evaluation of new SR products. Quarterly human landing catches will be done to assess the behavioral effects of the SR. The primary hypothesis on PE against the first-time malaria infection will be estimated by comparing the hazard rates of first-time malaria infection between SR and placebo upon the completion of the study in the ITT population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to <10 years
* Hb > 5mg/dl
* Sleeps in cluster >90% of nights during any given month
* No plans for extended travel (>1month) outside of home during study
* Not participating in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the Trial
* Provision of informed consent form signed by the parent(s) or guardian
* Children not on regular malaria prophylaxis° such as Proguanil
* Willingness to take AL and no history of hypersensitivity to AL

Exclusion Criteria:

* Children < 6 months or ≥ 10 years
* Hb ≤ 5 mg/dL, or Hb < 6mg/dL with signs of clinical decompensation
* Sleeps in cluster <90% of nights during any given month
* Plans for extended travel (>1month) outside of home during study
* Participating or planned participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure during the trial
* No provision of informed consent form signed by the parent(s) or guardian
* Children on regular malaria prophylaxis° such as Proguanil
* Unwillingness or refusal to take AL and history of AL hypersensitivity

  * Other malaria prophylaxis medicines: Mefloquine, Atavaquone/Proguanil (Malarone), Doxycycline, Tafenoquine, Sulfadoxine-Pyrimethamine (Fansidar), Amodiaquine and Co-trimoxazole (Septrin)

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5984 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
First-time malaria infection in core zones during intervention period. | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.

SECONDARY OUTCOMES:
Overall new malaria infections in core zones during intervention period. | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
Overall new malaria infections in buffer zones during intervention period. | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
Parasite-species-specific first-time malaria infections in the core zones. | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
Parasite-species-specific overall malaria infections in the core zones. | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
The first-time malaria infections in buffer zones during intervention period. | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
The first time malaria infections by two age groups (≤ 59 months old; 5 years to 10 years old). | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
Overall malaria infections by two age groups (≤ 59 months old; 5 years to 10 years old). | 12 months
  Measured by microscopy in children aged between 6 months to 10 years.
Anopheline-human contact (indoor and outdoor) using human biting rate (HBR) as an indicator for all anophelines and by anopheline species. | 12 months
  Measured by human-landing catch (HLC) during 12-h intervals on a quarterly basis during intervention period.
Anopheline parity rate as an indicator of population age structure for all anophelines and by anopheline species. | 12 months
  Measured by mosquito ovarian dissections from a sub-sample of anophelines collected during HLC procedures during intervention period.
Anopheline infectivity using sporozoite rate as an indicator for all anophelines and by anopheline species. | 12 months
  Measured by laboratory detection of sporozoites in mosquito head-preps from a sub-sample of anophelines collected during HLC and/or CDC-light trap procedures during intervention period.
Anopheline infectivity using EIR as an indicator for all anophelines and by anopheline species. | 12 months
  Measured by calculating the number of sporozoite-infected anopheline mosquitoes captured per person during intervention period from HLC and/or CDC-light trap procedures.
CDC-light trap indoor density for all anophelines and by anopheline species. | 12 months
  Measured by CDC-light trap collections during 12-h intervals on a monthly basis during intervention period.
Insecticide resistance. | 28 months
  Measured by WHO filter paper test and CDC bottle assays during baseline and intervention period.
Adverse Events and Serious Adverse Events. | 28 months
  Measured by solicited and unsolicited reports during baseline and intervention period. Mean, minimum and maximum frequency and percentage of AEs and SAEs across clusters among enrolled subjects will be summarized by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: John P Grieco, Ph.D., Study Director — University of Notre Dame; Eric Ochomo, Ph.D., Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Kenya (2):
  - Centers for Disease Control and Prevention, Busia, Busia County
  - Kenya Medical Research Institute (KEMRI), Busia, Busia County

IPD SHARING:
Plan to Share IPD: Yes
Analytical data will be anonymized and GPS tag-blurred to remove sensitive information prior to sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data and supporting information will be made available 12 months following completion of data analysis and will remain open access in the public domain.
Access Criteria: Open-access repository distributed under the terms of the Creative Commons Attribution (CC-BY) License, which permits unrestricted use, distribution, and reproduction in any medium, provided the original author and source are credited.

REFERENCES:
- [Background] Hamel MJ, Adazu K, Obor D, Sewe M, Vulule J, Williamson JM, Slutsker L, Feikin DR, Laserson KF. A reversal in reductions of child mortality in western Kenya, 2003-2009. Am J Trop Med Hyg. 2011 Oct;85(4):597-605. doi: 10.4269/ajtmh.2011.10-0678. PMID 21976557
- [Background] Zhou G, Afrane YA, Vardo-Zalik AM, Atieli H, Zhong D, Wamae P, Himeidan YE, Minakawa N, Githeko AK, Yan G. Changing patterns of malaria epidemiology between 2002 and 2010 in Western Kenya: the fall and rise of malaria. PLoS One. 2011;6(5):e20318. doi: 10.1371/journal.pone.0020318. Epub 2011 May 23. PMID 21629783
- [Background] Ogoma SB, Moore SJ, Maia MF. A systematic review of mosquito coils and passive emanators: defining recommendations for spatial repellency testing methodologies. Parasit Vectors. 2012 Dec 7;5:287. doi: 10.1186/1756-3305-5-287. PMID 23216844
- [Background] Ogoma SB, Ngonyani H, Simfukwe ET, Mseka A, Moore J, Killeen GF. Spatial repellency of transfluthrin-treated hessian strips against laboratory-reared Anopheles arabiensis mosquitoes in a semi-field tunnel cage. Parasit Vectors. 2012 Mar 20;5:54. doi: 10.1186/1756-3305-5-54. PMID 22433128
- [Background] Ogoma SB, Ngonyani H, Simfukwe ET, Mseka A, Moore J, Maia MF, Moore SJ, Lorenz LM. The mode of action of spatial repellents and their impact on vectorial capacity of Anopheles gambiae sensu stricto. PLoS One. 2014 Dec 8;9(12):e110433. doi: 10.1371/journal.pone.0110433. eCollection 2014. PMID 25485850
- [Background] Achee NL, Bangs MJ, Farlow R, Killeen GF, Lindsay S, Logan JG, Moore SJ, Rowland M, Sweeney K, Torr SJ, Zwiebel LJ, Grieco JP. Spatial repellents: from discovery and development to evidence-based validation. Malar J. 2012 May 14;11:164. doi: 10.1186/1475-2875-11-164. PMID 22583679
- [Background] Lucas JR, Shono Y, Iwasaki T, Ishiwatari T, Spero N, Benzon G. U.S. laboratory and field trials of metofluthrin (SumiOne) emanators for reducing mosquito biting outdoors. J Am Mosq Control Assoc. 2007 Mar;23(1):47-54. doi: 10.2987/8756-971X(2007)23[47:ULAFTO]2.0.CO;2. PMID 17536367
- [Background] Kawada H, Temu EA, Minjas JN, Matsumoto O, Iwasaki T, Takagi M. Field evaluation of spatial repellency of metofluthrin-impregnated plastic strips against Anopheles gambiae complex in Bagamoyo, coastal Tanzania. J Am Mosq Control Assoc. 2008 Sep;24(3):404-9. doi: 10.2987/5743.1. PMID 18939693
- [Background] Syafruddin D, Bangs MJ, Sidik D, Elyazar I, Asih PB, Chan K, Nurleila S, Nixon C, Hendarto J, Wahid I, Ishak H, Bogh C, Grieco JP, Achee NL, Baird JK. Impact of a spatial repellent on malaria incidence in two villages in Sumba, Indonesia. Am J Trop Med Hyg. 2014 Dec;91(6):1079-87. doi: 10.4269/ajtmh.13-0735. Epub 2014 Oct 13. PMID 25311699
- [Background] Hill N, Zhou HN, Wang P, Guo X, Carneiro I, Moore SJ. A household randomized, controlled trial of the efficacy of 0.03% transfluthrin coils alone and in combination with long-lasting insecticidal nets on the incidence of Plasmodium falciparum and Plasmodium vivax malaria in Western Yunnan Province, China. Malar J. 2014 May 31;13:208. doi: 10.1186/1475-2875-13-208. PMID 24885993
- [Derived] Ochomo EO, Gimnig JE, Awori Q, Abong'o B, Oria P, Ashitiba NK, Polo B, Moshi V, Otanga H, Adung'o F, Ouma EA, Outa S, Ramaita E, Levine R, Odongo W, Harvey SA, Monroe A, Hudson A, Sandberg B, Hendrickson J, Zhao X, Zhou R, Liu F, Achee NL, Grieco JP. Effect of a spatial repellent on malaria incidence in an area of western Kenya characterised by high malaria transmission, insecticide resistance, and universal coverage of insecticide treated nets (part of the AEGIS Consortium): a cluster-randomised, controlled trial. Lancet. 2025 Jan 11;405(10473):147-156. doi: 10.1016/S0140-6736(24)02253-0. Epub 2024 Dec 19. PMID 39709979
- [Derived] Ochomo EO, Gimnig JE, Bhattarai A, Samuels AM, Kariuki S, Okello G, Abong'o B, Ouma EA, Kosgei J, Munga S, Njagi K, Odongo W, Liu F, Grieco JP, Achee NL. Evaluation of the protective efficacy of a spatial repellent to reduce malaria incidence in children in western Kenya compared to placebo: study protocol for a cluster-randomized double-blinded control trial (the AEGIS program). Trials. 2022 Apr 5;23(1):260. doi: 10.1186/s13063-022-06196-x. PMID 35382858